CLINICAL TRIAL: NCT00007254
Title: Morphine-Infused Gel for Pressure Ulcer Analgesia
Brief Title: Morphine Gel for Bedsores
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR045506 (NIH); R01AR045506 (NIH); NIAMS-061
Record Dates: First submitted 2000-12-16; First posted 2000-12-18 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Decubitus Ulcer
Keywords: Analgesia; Bedsore; Morphine gel; Pressure ulcer; Pain; Ulcer
MeSH Terms: conditions — Pressure Ulcer; Agnosia; Pain; Ulcer | interventions — Analgesia

INTERVENTIONS:
Drug: Pain relief for pressure ulcers

SUMMARY:
This study tests the effectiveness of a morphine-containing gel for reducing pain caused by pressure ulcers, also known as bedsores or pressure sores. We will apply the gel containing morphine, or the gel alone, directly onto painful pressure ulcers and compare the results.

DETAILED DESCRIPTION:
In this study, we will apply a morphine-containing gel (or placebo) directly onto painful pressure ulcers. We will take participants off of any opioid-containing medications upon entry into the study. This allows us to measure any morphine that may enter into the bloodstream from the topically applied gel.

The purpose of this study is to examine the efficacy of the gel for pressure ulcer analgesia, as well as the systemic absorption of morphine from the topically applied gel. We will document the amount of pain medications taken by participants to determine whether the gel decreases the need for these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a Stage II pressure ulcer.
* Pressure ulcer must be painful.
* Primary Care physician must approve participation.
* Thinking ability must be clear and intact.
* Willing to change pain medication to oxycodone.

Exclusion Criteria:

* Allergy to morphine, oxycodone or intrasite gel.
* Use of codeine- or morphine-containing medications.
* Use of pain medications for anything other than the pressure ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2000-03; Study Completion 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Teresa D. Long, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Kindred Hospital, Kansas City, Missouri

REFERENCES:
- [Background] Twillman RK, Long TD, Cathers TA, Mueller DW. Treatment of painful skin ulcers with topical opioids. J Pain Symptom Manage. 1999 Apr;17(4):288-92. doi: 10.1016/s0885-3924(98)00140-7. PMID 10203881